CLINICAL TRIAL: NCT07306533
Title: Effect of Menstrual Phase on the Anesthetic Efficacy of Inferior Alveolar Nerve Block in Patients With Symptomatic Irreversible Pulpitis in Mandibular Molars
Brief Title: Effect of Menstrual Phase on the Anesthetic Efficacy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jamia Millia Islamia (Other)
Responsible Party: Principal Investigator, Dr. Vivek Aggarwal, Professor, Jamia Millia Islamia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Menstrual Phase
Record Dates: First submitted 2025-12-12; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Pulpitis - Irreversible
Keywords: IANB; pulpitis; anesthesia
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inferior Alveolar Nerve Block (Experimental): Patients will receive a standard inferior alveolar nerve block using 1.5 mL of 2% lidocaine with 1:80,000 epinephrine. The efficacy of anesthesia will be evaluated by two measures. First, pulpal anesthesia will be assessed using a cold test with Endo-Ice. Second, intraoperative pain will be recorded during access cavity preparation using the Heft-Parker Visual Analog Scale (HPVAS). Anesthetic outcome will be classified as either success or failure. Success will be defined as absence of response to cold testing along with no or only mild intraoperative pain (HPVAS ≤ 54 mm).
  Interventions: Procedure: Inferior Alveolar Nerve Block

INTERVENTIONS:
Procedure: Inferior Alveolar Nerve Block — The patients will receive a standard inferior alveolar nerve block using 1.5 mL of 2% lidocaine with 1:80,000 epinephrine. The efficacy of anesthesia will be evaluated by two measures. First, pulpal anesthesia will be assessed using a cold test with Endo-Ice. Second, intraoperative pain will be recorded during access cavity preparation using the Heft-Parker Visual Analog Scale (HPVAS). Anesthetic outcome will be classified as either success or failure. Success will be defined as absence of response to cold testing along with no or only mild intraoperative pain (HPVAS ≤ 54 mm).

SUMMARY:
The goal of this observational prospective clinical study is to learn whether the menstrual phase influences the anesthetic efficacy of inferior alveolar nerve block (IANB) in female patients aged 20-40 years with symptomatic irreversible pulpitis in mandibular molars. The main questions it aims to answer are:

Does the success rate of IANB vary across different phases of the menstrual cycle?

Are certain menstrual phases associated with a higher likelihood of anesthetic failure during endodontic access preparation?

Researchers will compare five menstrual phase groups (menstrual, follicular, ovulatory, luteal, and premenstrual) to see if hormonal fluctuations affect anesthetic success.

Participants will:

Receive a standardized inferior alveolar nerve block using 2% lidocaine with 1:80,000 epinephrine

Undergo cold testing and access cavity preparation to assess anesthetic success

Have intraoperative pain recorded using the Heft-Parker Visual Analog Scale (HPVAS), with menstrual phase information recorded confidentially and blinded to the treating clinician

DETAILED DESCRIPTION:
Introduction Pain management is fundamental to the success of dental procedures, particularly in endodontics, where patients often present with severe preoperative pain due to irreversible pulpitis. The inferior alveolar nerve block (IANB) is the most frequently employed anesthetic technique for mandibular molars, yet its reliability in inflamed pulpal conditions remains questionable. Numerous studies have documented variable efficacy, with failure rates ranging between 30% and 80%, despite correct technique and the use of appropriate anesthetic agents (1). This unpredictability poses a significant challenge, often necessitating supplemental injections such as intraligamentary, intraosseous, or intrapulpal techniques to achieve adequate pain control.

Traditionally, the reasons for IANB failure in irreversible pulpitis have been attributed to local and central mechanisms. Locally, inflammation-induced acidosis decreases the proportion of anesthetic molecules in their non-ionized, membrane-penetrating form, thereby reducing nerve blockade efficiency (2). Inflammatory mediators, including prostaglandins and bradykinin, also sensitize nociceptors and increase expression of tetrodotoxin-resistant sodium channels, which are inherently less sensitive to lidocaine and other amide anesthetics. At the central level, hyperalgesia and central sensitization amplify nociceptive transmission, contributing to anesthetic resistance (1). Patient-related variables, such as anxiety and fear, further modulate pain perception and anesthetic outcome.

However, even after controlling for these factors, considerable inter-individual variability remains unexplained, suggesting a systemic or constitutional influence. Increasing attention has therefore been directed toward genetic, hormonal, and gender-related factors as potential modulators of anesthetic efficacy.

A large body of literature has established sex-based differences in pain perception. Women consistently report a higher prevalence of pain conditions such as migraine, temporomandibular disorders, and fibromyalgia compared to men (3). Experimental models demonstrate that women often have lower pain thresholds, reduced tolerance to noxious stimuli, and enhanced temporal summation of pain (4). These findings suggest an inherent biological variability in nociceptive processing, which extends to the clinical response to local anesthesia. Indeed, several dental anesthesia studies have observed that women require supplemental injections more frequently than men for comparable procedures (Aggarwal et al., 2009).The underlying mechanism for these sex differences is multifactorial. While psychological and cultural factors may influence pain reporting, biological variables-particularly the role of sex hormones-are now considered central.

The menstrual cycle is characterized by cyclical fluctuations in estrogen and progesterone. These hormones exert significant effects on nociceptive transmission and pain perception at peripheral, spinal, and supraspinal levels.Estrogen has dual, context-dependent effects. It can enhance excitability of nociceptive neurons by upregulating sodium channels and NMDA receptors, thereby facilitating pain (4). Conversely, estrogen also promotes endogenous opioid activity, especially via μ-opioid receptors in the central nervous system, which can increase pain inhibition (5).Progesterone is thought to lower pain thresholds by modulating GABAergic and sodium channel activity. High-progesterone phases, such as the luteal and premenstrual phases, have been associated with increased sensitivity to painful stimuli (4, 5).

Together, these hormonal fluctuations create a dynamic pain response across the menstrual cycle. For example, studies have reported that tolerance to electrical pain stimulation is higher in the luteal phase, while sensitivity to thermal and mechanical pain is increased during the same period (4-6).

Although medical and dental literature directly linking menstrual phases to anesthetic outcomes is limited, there is indirect evidence to suggest such an association. In obstetric anesthesia, variable efficacy of epidural and spinal anesthesia has been reported at different stages of the menstrual cycle, attributed to hormonal modulation of sodium channels and opioid receptor sensitivity (4). In dentistry, anecdotal clinical observations and limited studies suggest that female patients may exhibit reduced anesthetic efficacy during luteal and premenstrual phases, when progesterone levels peak.

Rationale for the Present Study: Given the high prevalence of IANB failure in irreversible pulpitis and the underexplored role of menstrual cycle phases, there is a clear need to systematically investigate this association. Most current anesthetic strategies do not account for hormonal influences, yet understanding these variations could provide a scientific basis for predicting anesthetic efficacy and improving pain management in female patients. By evaluating the success of IANB in different menstrual phases, this study seeks to fill an important gap in dental anesthesia research and contribute to personalized approaches in endodontics.

Aims and Objectives Primary Aim To evaluate the association between menstrual phase and the clinical success rate of IANB in mandibular molars with irreversible pulpitis.

Objectives

1. To categorize patients according to their menstrual cycle phase.
2. To assess anesthetic success following IANB during each menstrual phase.
3. To compare success rates across phases to identify significant differences.
4. To analyze the potential role of hormonal fluctuations as predictors of anesthetic efficacy.

Materials and Methods Study Design: Observational prospective clinical study. Study Population: Female patients aged 20-40 years presenting with symptomatic irreversible pulpitis in mandibular first or second molars.

Grouping

Patients will be divided into five groups based on menstrual cycle phase (day 1 = first day of menstruation):

* Menstrual: Days 1-5
* Follicular: Days 6-12
* Ovulatory: Days 13-16
* Luteal: Days 17-23
* Premenstrual: Days 24-28 (Self-reported menstrual phase will be cross-checked with cycle history. Information will remain blinded to the treating clinician.) Intervention All patients enrolled in the study will receive a standard inferior alveolar nerve block using 1.5 mL of 2% lidocaine with 1:80,000 epinephrine. The efficacy of anesthesia will be evaluated by two measures. First, pulpal anesthesia will be assessed using a cold test with Endo-Ice. Second, intraoperative pain will be recorded during access cavity preparation using the Heft-Parker Visual Analog Scale (HPVAS). Anesthetic outcome will be classified as either success or failure. Success will be defined as absence of response to cold testing along with no or only mild intraoperative pain (HPVAS ≤ 54 mm). Failure will be recorded when patients exhibit a positive cold test response and/or report moderate to severe intraoperative pain (HPVAS > 54 mm) despite IANB administration.

Sample Size Calculation Assuming an expected difference of ~30% in anesthetic success between phases, with 80% power and 5% significance, minimum 30 patients per group are required. Total sample size: 150 patients.

Statistical Analysis All collected data will first be subjected to descriptive statistical analysis to summarize demographic characteristics such as age distribution and baseline pain scores across the study groups. The association between menstrual phase and the success rate of inferior alveolar nerve block will be evaluated using the chi-square test. To further account for potential confounding variables, including age and baseline preoperative pain intensity, logistic regression analysis will be performed. Statistical significance will be set at a p-value of less than 0.05.

Work Schedule The estimated duration of the study is nine months. The initial six months will be devoted to recruitment of eligible participants and collection of clinical and outcome data. This will be followed by a three-month period dedicated to data analysis, statistical interpretation, and preparation of the study report and manuscript.

ELIGIBILITY:
Inclusion Criteria

* Female patients aged 20-40 years.
* Regular menstrual cycles (28 ± 3 days).
* Diagnosed with symptomatic irreversible pulpitis in mandibular molars.
* Indicated for root canal therapy.
* Willing to provide informed consent. Exclusion Criteria
* Use of oral contraceptives or hormonal therapy.
* Irregular menstrual cycles.
* Pregnancy or lactation.
* Systemic disease affecting pain perception (e.g., diabetes, neuropathies).
* Recent use of analgesics or sedatives (within 24 hours).
* Allergy to local anesthetics.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Mensturating females
Enrollment: 150 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Anesthetic success | From enrollment to the end of treatment at 10 months, success will be evaluated after 5 minutes of administrtion if IANB.
  The efficacy of anesthesia will be evaluated by two measures. First, pulpal anesthesia will be assessed using a cold test with Endo-Ice. Second, intraoperative pain will be recorded during access cavity preparation using the Heft-Parker Visual Analog Scale (HPVAS). Anesthetic outcome will be classified as either success or failure. Success will be defined as absence of response to cold testing along with no or only mild intraoperative pain (HPVAS ≤ 54 mm). Failure will be recorded when patients exhibit a positive cold test response and/or report moderate to severe intraoperative pain (HPVAS > 54 mm) despite IANB administration.
Intraoperative pain | From enrollment to the end of treatment at 10 months, success will be evaluated during the treatment.
  The intraoperative pain shall be measured using a 170mm HP visual anlouge scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, JMI, New Delhi, Delhi(दिल्ली), India

IPD SHARING:
Plan to Share IPD: Yes
The data collected in this study will be used solely for the purposes outlined in the approved research protocol and for publication in aggregated, anonymized form, without any identifiers that could reveal individual participant information.
Supporting Information: Study Protocol
Time Frame: After 1 year of completion of study